CLINICAL TRIAL: NCT01447368
Title: Comparison of Medical Therapy (Oral Cinacalcet) Versus Surgical Therapy (Total Parathyroidectomy) on Vascular/Valvular Calcification in Chronic Peritoneal Dialysis Patients With Secondary Hyperparathyroidism - A Pilot Randomized Study
Brief Title: Cinacalcet Versus Parathyroidectomy in Peritoneal Dialysis Patients
Acronym: PROCEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Honorary Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-2015
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Kidney Failure; Secondary Hyperparathyroidism; Vascular Diseases
Keywords: chronic kidney disease; peritoneal dialysis; secondary hyperparathyroidism; parathyroidectomy; vascular calcification; cinacalcet
MeSH Terms: conditions — Renal Insufficiency; Hyperparathyroidism, Secondary; Vascular Diseases; Renal Insufficiency, Chronic; Vascular Calcification | interventions — Cinacalcet

STUDY DESIGN:
Intervention Model Description: Cinacalcet medical treatment versus total parathyroidectomy with forearm autografting surgical treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cinacalcet treatment (Experimental): Oral Cinacalcet treatment arm, 25mg daily to be administered and gradually step up as required to control iPTH between 2 - 9 times lab reference range, Maximum dose to be given is 100mg daily
  Interventions: Drug: Cinacalcet
- Surgical total parathyroidectomy (Active Comparator): Surgical total parathyroidectomy with forearm autografting will be performed for patients randomized to this arm.
  Interventions: Procedure: Surgical total parathyroidectomy with forearm autografting

INTERVENTIONS:
Drug: Cinacalcet — oral cinacalcet 25mg once daily as a start and up titrated by 25mg daily according to response in lowering PTH and maximum oral dose allowed is 100mg daily
  Other Names: Regpara
  Arms: Cinacalcet treatment
Procedure: Surgical total parathyroidectomy with forearm autografting — Surgical total parathyroidectomy with forearm autografting will be performed
  Arms: Surgical total parathyroidectomy

SUMMARY:
This is a pilot, prospective randomized controlled study with the primary objective to evaluate and compare medical treatment of severe SHPT, namely oral cinacalcet versus surgical treatment, that is, parathyroidectomy with forearm autografting, on the progression of coronary artery and valvular calcification and left ventricular mass index in endstage renal disease patients receiving peritoneal dialysis over 12 months. The change in arterial stiffening, left ventricular volume, aortic valve calcium score and bone mineral density, nutritional status and biochemical parameters, quality of life measures will be evaluated as secondary objectives of this study.

DETAILED DESCRIPTION:
Patients with severe secondary hyperparathyroidism (SHPT) are frequently complicated with vascular calcification. There is some suggestion that subtotal parathyroidectomy may reduce or stabilize vascular calcium scores in dialysis patients. Experimental data suggests that SHPT plays an important role in mediating uraemic arterial disease and that parathyroidectomy largely prevented the development of calcification. Cinacalcet has emerged as a novel therapy for the treatment of SHPT and has been shown to reduce the need for surgical parathyroidectomy. However, their effects on vascular, cardiac, bone and nutrition status have not been evaluated and compared with parathyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ESRD patients on long-term peritoneal dialysis treatment, with elevated intact parathyroid hormone (iPTH) levels > 800pg/mL.
2. Patients with parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan.
3. Patients with age between 18 - 75 years.

Exclusion Criteria:

1. Patients with background valvular heart disease
2. Patients who are unfit for general anaesthesia
3. Patients with acute myocardial infarction within recent two months
4. Patients with poor general condition
5. Patients with plans for living related kidney transplant within 1 year
6. Patients with previous history of parathyroidectomy
7. Patients with underlying malignancy
8. Patients with hepatic dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-05-10 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Change in coronary artery calcium score | 52 weeks
  Change in coronary artery calcium score
change in left ventricular mass index | 52 weeks
  change in left ventricular mass index

SECONDARY OUTCOMES:
change in left ventricular volume and ejection fraction | 52 weeks
  change in left ventricular volume and ejection fraction
Change in aortic pulse wave velocity | 24 and 52 weeks
  Change in aortic pulse wave velocity
Change in aortic valve and mitral valve calcium score | 52 weeks
  Change in aortic valve and mitral valve calcium score
change in augmentation index and heart rate adjusted augmentation index | over 52 weeks
  change in augmentation index and heart rate adjusted augmentation index
change in bone mineral density at forearm, spine and femur | 52 weeks
  change in bone mineral density at forearm, spine and femur
Quality of Life (QOL) scores | 52 weeks
  Kidney Disease Outcome Quality Initiatives (KDOQI QOL domain scores)
change in resting energy expenditure | 24 and 52 weeks
  Change in resting energy expenditure
change in lean muscle mass | 52 weeks
  Change in lean muscle mass
change in handgrip strength | 24 and 52 weeks
  Change in handgrip strength
Change in subjective global assessment | 24 and 52 weeks
  Change in subjective global assessment
Change in serum calcium and phosphorus | over 52 weeks
  Change in biochemical parameter Serum calcium and phosphorus
change in intact parathyroid hormone (iPTH) level | 52 weeks
  Change in biochemical parameter Parathyroid hormone
Change in alkaline phosphatase | over 52 weeks
  Change in biochemical parameter alkaline phosphatase
change in serum albumin | over 52 weeks
  CHange in biochemical parameter serum albumin
change in lymphocyte count | over 52 weeks
  change in lymphocyte count
change in lipid profile | over 52 weeks
  change in lipid profile
change in systolic and diastolic blood pressure | over 52 weeks
  change in systolic and diastolic blood pressure
change in subendocardial viability ratio | over 52 weeks
  change in subendocardial viability ratio

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, PhD, Principal Investigator — University of Hong Kong, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital and Tung Wah Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang AY, Tang TK, Yau YY, Lo WK. Impact of Parathyroidectomy Versus Oral Cinacalcet on Bone Mineral Density in Patients on Peritoneal Dialysis With Advanced Secondary Hyperparathyroidism: The PROCEED Pilot Randomized Trial. Am J Kidney Dis. 2024 Apr;83(4):456-466.e1. doi: 10.1053/j.ajkd.2023.10.007. Epub 2023 Nov 30. PMID 38040277
- [Derived] Wang AY, Lo WK, Cheung SC, Tang TK, Yau YY, Lang BH. Parathyroidectomy versus oral cinacalcet on cardiovascular parameters in peritoneal dialysis patients with advanced secondary hyperparathyroidism (PROCEED): a randomized trial. Nephrol Dial Transplant. 2023 Jul 31;38(8):1823-1835. doi: 10.1093/ndt/gfad043. PMID 36869794